CLINICAL TRIAL: NCT05415891
Title: Improving the Integration of Mental Health and Substance Use Treatment Into Ryan White-Funded Care Sites in Atlanta Using an Implementation Science Approach
Brief Title: The IMPROV Project: Improving Mental Health and Substance Use Treatment Provision (IMPROV) Among People Living With HIV (Human Immunodeficiency Virus) in Atlanta
Acronym: IMPROV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RTI International (Other)
Collaborators: SisterLove, Inc. (Other Government); Positive Impact Health Centers (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00063322; R34MH124628 (NIH)
Record Dates: First submitted 2022-06-08; First posted 2022-06-13 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Mental Health Disorder; Substance Use Disorder; Stigmatization; Implementation Science
Keywords: Mental Health Disorder; Substance use Disorder; Human Immunodeficiency Virus; Comorbidity; Treatment; Implementation Science
MeSH Terms: conditions — Mental Disorders; Substance-Related Disorders; Stereotyping; Acquired Immunodeficiency Syndrome | interventions — N-(4'-fluorobutyrophenone)-4-(4-chlorophenyl)pyridinium

STUDY DESIGN:
Intervention Model Description: This study will include two levels of randomization: clinic level and provider level. We will randomize the two clinic study sites into one of two study conditions. One clinic will be randomized to the stigma-reduction training arm, and one clinic will be randomized to the no stigma-reduction training arm (but will receive the training at the end of the study). At the provider level, we will use a multiple baseline design that is fundamental to idiographic approaches. All providers will receive the You℞ Decision prescribing platform. Providers will be randomized to one of four intervention schedules: (a) 1-week baseline + 11-week intervention, (b) 2-week baseline + 10-week intervention, (c) 3-week baseline + 9-week intervention, and (d) 4-week baseline + 8-week intervention. Randomization will be stratified by clinic. Two providers (one from each site) will be randomized to each intervention schedule (for a total of 8 providers).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stigma-Reduction Training Arm + YouRx Prescribing Platform (Experimental): Staff working in the clinic in this arm will be offered a whole-site stigma reduction training.
  Participating HIV care providers will have access to the YouRx Prescribing Platform.
  Interventions: Behavioral: Modified Health Policy Project (HPP) HIV-Stigma and Discrimination Reduction Training Curriculum; Device: You℞ Decision prescribing platform
- YouRx Prescribing Platform Only (Experimental): Staff working in the clinic in this arm will not be offered a whole-site stigma reduction training. However, staff will be offered this training at the conclusion of the study.
  Participating HIV care providers will have access to the YouRx Prescribing Platform.
  Interventions: Device: You℞ Decision prescribing platform

INTERVENTIONS:
Behavioral: Modified Health Policy Project (HPP) HIV-Stigma and Discrimination Reduction Training Curriculum — The Health Policy Project (HPP) training curriculum provides participatory training modules that address three key actionable drivers of HIV-stigma. The HPP curriculum was adapted through participatory workshops with the study's community collaborative board, including representatives from the HIV care and advocacy communities as well as community members. The training is a whole-site training to address stigma as a barrier to accessing substance use and mental health services by persons living with HIV. Consequently, staff at all levels (clinical and nonclinical) will be trained on stigma and discrimination as it relates to persons living with HIV in order to reduce stigma-related barriers to mental health and substance use healthcare in Positive Impact Health Centers and increase retention in healthcare services for persons living with HIV.
  Arms: Stigma-Reduction Training Arm + YouRx Prescribing Platform
Device: You℞ Decision prescribing platform — The You℞ Decision prescribing platform is a mobile application that serves as a reference to quickly inform providers about the medications recommended for serious mental health disorders and naltrexone to treat AUD; the appropriate dosing regimen; and potential contraindications or interactions related to antiretroviral therapy medications or other psychiatric medication. Information for the platform is adapted from the Department of Veteran Affairs' Manual for HIV Care in Primary Care settings.

SUMMARY:
This project consists of a pilot trial to assess the preliminary impact of a stigma-reduction training to reduce clinic-level stigma and the You℞ Decision prescribing platform to increase HIV care providers' self-efficacy related to prescribing psychiatric medication for depression, post-traumatic stress disorder (PTSD), and bipolar disorder as well as naltrexone for alcohol use disorder (AUD).

DETAILED DESCRIPTION:
The study will pilot test a two-level strategy to improve integration of pharmacotherapy for serious mental health and alcohol use disorders among people living with HIV (PLHIV) in Ryan White-funded healthcare centers in Atlanta, Georgia. A small pilot trial will be conducted in the two clinic study sites to assess the acceptability, feasibility, adoption, and preliminary impact of a stigma-reduction training and the You℞ Decision prescribing platform.

The researchers will fulfill the purpose of this study through the following aims:

Aim 1: To conduct formative activities with PLHIV, HIV care providers, and our Community Collaborative Board (CCB) to adapt a stigma-reduction training to address mental health and substance abuse-related stigma among clinic staff and engage HIV care providers and an expert panel to develop the You℞ Decision prescribing platform to support HIV care providers to offer pharmacotherapy to treat depression, PTSD, bipolar disorder, and AUD (completed).

Aim 2: To assess the acceptability of the stigma-reduction training among clinic staff and the feasibility, acceptability, and adoption of the You℞ Decision prescribing platform during clinical encounters among providers in HIV care settings.

Aim 3: To use idiographic methods to conduct a pilot trial to assess the preliminary impact of the stigma-reduction training on clinic-level stigma and of the You℞ Decision prescribing platform on HIV care providers' self-efficacy to prescribe psychiatric medications and naltrexone as well as the impact of the stigma-reduction training and platform to increase the percentage of eligible patients who receive and accept prescriptions to treat depression, PTSD, bipolar disorder, and AUD.

This implementation science study aims to reduce HIV-associated comorbidities by improving the integration of mental health and AUD treatment into Ryan White-funded care sites. If the findings indicate that the stigma-reduction training and prescribing platform are feasible, this study will be the impetus for the scale up these strategies to additional Ryan White-funded care sites in Georgia.

ELIGIBILITY:
Inclusion Criteria:

Stigma Reduction Training

* be 18 years of age or older
* be a staff member at the clinic study site randomized for the stigma-reduction training

Clinic Staff Survey

* work at one of the two clinic study sites
* be 18 years of age or older

Patient Survey

* 18 or older
* report being HIV positive
* have received care from a clinic study site recently

Pilot Trial

* provide HIV care
* be 18 years of age or older
* be licensed to provide prescription medication
* provide care at one of the two clinic study sites

Exclusion Criteria:

Stigma Reduction Training

* Have been part of the formative activities

Clinic Staff Survey

* Have been part of the formative activities.

Patient Survey

* HIV negative
* Have not attended a study clinic site recently
* Have participated in the formative activities

Pilot Trial

* Not a prescribing provider
* Not a provider at a study clinic site recently
* Have been part of the formative activities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 333 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Clinic Staff-Level Outcome: Acceptability of Stigma Reduction Training | Immediately post-training
  4-item self-report measure to assess clinic staff's satisfaction with the stigma reduction training
Provider-Level Outcome: Acceptability of the YouRx Decision Prescribing Platform | 3 months follow-up
  4-item measure to assess provider satisfaction with the You℞ Decision platform
Provider-Level Outcome: Feasibility of the YouRx Decision Prescribing Platform | 3 months follow-up
  4-item measure to assess provider perception that the You℞ Decision platform can be integrated into usual care
Provider-Level Outcome: Adoption of the YouRx Decision Prescribing Platform | Weekly (12 weeks)
  Provider use of the You℞ Decision prescribing platform
Provider-Level Outcome: Usability of the YouRx Decision Prescribing Platform | 3 months follow-up
  21-item survey to assess the ease of use of the You℞ Decision prescribing platform
Clinic Staff-Level Outcome: Observed Stigma Reduction | 3 months follow-up
  Clinic staff observed stigmatizing behaviors toward those with serious mental health and/or substance use disorders
Health Consumer-Level Outcome: Observed Stigma Reduction | 3 months follow-up
  Experienced or observed stigma and discrimination from clinic staff based on serious mental health or substance use disorder
Provider-Level Outcome: Provider Self-Efficacy | 3 months follow-up
  11-item survey to assess providers confidence to treat serious mental health disorders and AUD
Clinic-Level Outcome: Adoption of Psychiatric Medication and Naltrexone | 3 months follow-up
  Percentage of eligible patients who receive a prescription for psychiatric medication or naltrexone or an in-house referral for psychiatric treatment from their HIV care provider.
Clinic-Level Outcome: Reach of Prescription of Psychiatric Medication and Naltrexone | 3 months follow-up
  Percentage of eligible patients who fulfill a prescription for a psychiatric medication or naltrexone or in-house referrals at the clinic level
  Percentage of eligible patients who fill a prescription for psychiatric medication or naltrexone or attend an intake appointment with an in-house mental health or substance use provider.

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Peasant Bonner, PhD, Principal Investigator — RTI International
Locations (2):
- United States (2):
  - Positive Impact Health Center--Decatur Location, Decatur, Georgia
  - Positive Impact Health Center--Duluth Location, Duluth, Georgia

IPD SHARING:
Plan to Share IPD: No